CLINICAL TRIAL: NCT03069053
Title: Clinical Features and Histologic Findings in Bladder Pain Syndrome/Interstitial Cystitis (BPS/IS): New Findings on Useful Correlations
Brief Title: Clinical Features and Histologic Findings in Bladder Pain Syndrome/Interstitial Cystitis
Acronym: HistologyIC
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Daniele Porru, Principal Invesigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: IRCCSPSMATTEO
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Interstitial Cystitis, Chronic; Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Biospecimen Retention: Samples Without DNA — bladder biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives- to find out whether a correlation exists between denudation of urothelium and diagnosic delay in patients with BPS / IC, secondary aim was to search a correlation between impact of symptoms evaluated with ICSI-ICPI and number of comorbid conditions associated with BPS-IC.

Patients and Methods- Fifty-seven consecutive patients underwent cystoscopy under anaesthesia to classify those cases suspected of BPS/IC. As for the evaluation of the ICSI-ICPI scores we considered significant relevant values those ≥ 12. Patients underwent cystoscopy with hydrodistension under general (90%) or locoregional anaesthesia. Bladder biopsies were taken, including detrusor muscle, from those areas with the most apparent bladder wall lesions. All biopsies were then fixed in 4% formalin and sent to the Pathologist for examination.

DETAILED DESCRIPTION:
Between 2005 and 2016, in our Department 57 consecutive patients underwent cystoscopy under anaesthesia to classify those cases suspected of BPS/IC. Patients reported long-lasting irritative bladder symptoms, including urgency, daytime frequency of seven or more episodes, nocturia, and pain in the lower abdomen, lower back, vagina or perineum during filling or after micturition. Alternative diagnoses such as urinary tract infection (UTI) were excluded. Confusable diseases were ruled out by thorough history, clinical examination, urine analysis and imaging.

By means of a detailed medical history we considered the time of symptom onset, frequency of micturitions, the presence of associated diseases. All patients were given the same questionnaire (O'Leary-Sant Interstitial Cystitis Symptom and Problem Index) (19), filled at the time of bladder biopsy.

As for the evaluation of the ICSI-ICPI scores we considered significant relevant values those ≥ 12.

All patients underwent cystoscopy with hydrodistension under general (90%) or locoregional anaesthesia. A rigid cystoscope with a Ch. 22 caliber was used, mannitol solution was used as filling fluid, and infusion height was 80 cm above the symphysis pubis. During filling the bladder was continuously inspected. At maximal capacity, distension was maintained until spontaneous filling stopped and maximum capacity was reached. At this point the bladder was drained and bladder walls and mucosa were closely examined . The bladder was then filled again at approximately half capacity, and at least three deep biopsies were taken, including detrusor muscle, from those areas with the most apparent bladder wall lesions.

All biopsies were then fixed in 4% formalin and sent to the Pathologist for examination. It was specifically asked to assess the presence of urothelial denudation, inflammatory infiltrate, counts of mast cells in the submucosa and detrusor, presence of intrafascicular fibrosis and submucosal bleeding. A cut-off of 28 mast cells / mm2 was used for the assessment of detrusor mastocytosis.

Morphologic Study Biopsy samples were cut in 5-μm-thick sections, then stained with the following reagents for morphologic evaluation: Hematoxylin-Eosin, Giemsa and Masson Tricromic Stain. This procedure was performed by automatic stainers (Leica, mod. ST5020 and mod. Autostainer™ XL).

In each biopsy the following parameters were evaluated, according to the recommendations reported by Hanno et al. (20) and reported in Table 1.

If the biopsy wasn't adequately sized (< 1 mm2-wide), we decided to evaluate the most reliable parameters, giving a N.V. (Not Valuable) response to the others.

Such parameters were single-blindly studied by two independent pathologists using optic microscopes (Nikon, mod. Eclipse™ E400 and mod. Eclipse™ CI) and discordant cases were then discussed jointly.

Immunohistochemical Studies Immunohistochemical reactions with Dako monoclonal antibody anti-Human Mast-cell Tryptase (Clone AA1; IgG1, Kappa), at 1:4000 dilution, were performed in order to highlight the mast-cell component of the inflammatory infiltrate, and then to quantify it. According to the protocol followed at the Laboratory of Immunohistochemistry of the Pathology Unit the automatic immunostainer Dako Omnis™ was used.

Evaluation of the Immunostainings

The reactions were evaluated using optic microscopes (Nikon, mod. Eclipse™ E400 and mod. Eclipse™ CI). The following parameters were studied:

* Number of mast-cells/mm2 of mucosa;
* Number of mast-cells/mm2 of submucosa;
* Number of mast-cells/mm2 of the detrusor layer. In order to obtain the highest accuracy, a single-blind evaluation was performed by two independent pathologists; discordant or uncertain cases were then discussed jointly.

All patients were evaluated retrospectively using patient files, they were given a score between 0 to 5 according to the presence of the following criteria (each criteria counting one point): pain, nocturia, a bladder capacity of 500 mL, glomerulations, or interfascicular fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients reported long-lasting irritative bladder symptoms, including urgency, daytime frequency of seven or more episodes, nocturia, and pain in the lower abdomen, lower back, vagina or perineum during filling or after micturition.

Exclusion Criteria:

* Alternative diagnoses such as urinary tract infection (UTI) were excluded. Confusable diseases were ruled out by thorough history, clinical examination, urine analysis and imaging.

Ages: 19 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty-seven consecutive patients underwent cystoscopy under anaesthesia to classify those cases suspected of BPS/IC
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
correlation between denudation of urothelium and diagnosic delay | 11 years
  to find out whether a correlation exists between denudation of urothelium and diagnosic delay in patients with BPS / IC

SECONDARY OUTCOMES:
correlation between impact of symptoms evaluated with ICSI-ICPI and number of comorbid conditions associated with IC | 11 years
  to search a correlation between impact of symptoms evaluated with ICSI-ICPI and number of comorbid conditions associated with IC

CONTACTS AND LOCATIONS:
Overall Officials: DANIELE PORRU, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
Locations (4):
- Italy (4):
  - Clinical Epidemiology and Biometric Unit, Fondazione IRCCS Policlinico San Matteo, Pavia
  - Histology and Pathology Service, Fondazione IRCCS Policlinico San Matteo, Pavia
  - Obstetric and Gynecological Clinic, Fondazione IRCCS Policlinico San Matteo, Pavia
  - Urology Department Fondazione IRCCS Policlinico San Matteo, Pavia

IPD SHARING:
Plan to Share IPD: No